CLINICAL TRIAL: NCT04069052
Title: The Effect of Inhaled Nitric Oxide (iNO) on Physiologic Dead Space in Patients With Mild Chronic Obstructive Pulmonary Disease
Brief Title: The Effect of Inhaled Nitric Oxide on Deadspace in COPD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dr. Denis O'Donnell (Other)
Responsible Party: Sponsor-Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DMED-2274-19
Record Dates: First submitted 2019-07-11; First posted 2019-08-28 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Dyspnea; Exertional Dyspnea; Dead Space; Exercise; Inspiratory Neural Drive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity | interventions — Nitric Oxide

STUDY DESIGN:
Intervention Model Description: Single-centre, double-blinded, crossover study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled Nitric Oxide (Experimental): Inhaled nitric oxide administered throughout 4 min exercise protocol at 800 ppm.
  Interventions: Drug: Nitric Oxide
- Placebo (Placebo Comparator): Inhaled room air administered throughout 4 min exercise protocol at FiO2 = 0.21.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitric Oxide — Gaseous pulmonary vasodilator, SoKinox (nitric oxide) flowed into a mask and breathed in.
  Other Names: SoKinox
  Arms: Inhaled Nitric Oxide
Drug: Placebo — Room air (placebo) flowed into a mask and breathed in.
  Other Names: Room air
  Arms: Placebo

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a progressive disease of the respiratory system that generally develops as a result of smoking. Most people with COPD are classified as having "mild" disease severity and may not have significantly impaired lung function (e.g. flow) as measured by traditional lung function tests. However, multiple studies have shown that patients with mild disease already have significant damage to the small airways and blood vessels of the pulmonary system. This results in a considerable portion of the lung that does not participate in gas exchange, a phenomenon called physiologic dead space. Mild COPD patients develop symptoms of intolerable breathlessness early in exercise compared with healthy individuals. Previous studies have shown that pulmonary vasodilators, which locally increase blood vessel radius, may improve gas exchange and reduce symptoms of breathlessness in patients with mild COPD. Therefore, the objective of this study is to determine the effect of reducing dead space with a pulmonary vasodilator on the intensity of breathlessness during exercise in patients with mild COPD. This five visit, double-blinded, placebo-controlled crossover study will test the impact of inhaled nitric oxide, a direct vasodilator, during cardiopulmonary exercise on dead space and breathlessness intensity. Use of an esophageal catheter during testing will additionally permit measurement of neural drive to breathe and pulmonary mechanics throughout the protocol. Though patients with mild COPD represent the majority of the COPD population, their symptoms remain poorly managed by current, inefficient standard of care. The proposed study will examine dead space reduction as a novel therapeutic target for improving breathlessness and exercise tolerance in patients with mild COPD.

DETAILED DESCRIPTION:
This study will recruit 20 current or ex-smokers who meet the criteria for mild chronic obstructive pulmonary disease (COPD), measured by lung function tests. Participation is voluntary and participants may withdraw from the study at any time.

Procedures:

General Medical Examination: All participants will undergo a physical examination conducted by a physician. Concomitant medications will be recorded as well as body height and weight; blood pressure; heart rate rhythm using a 12-lead electrocardiogram (ECG); and blood oxygen saturation. The physician will identify any contraindications to exercise testing that would prevent safe participation.

Pulmonary Function Tests: Standard lung function tests include: spirometry (measuring respiratory flow during a maximal breath outward); body plethysmography (measuring lung volumes); diffusing capacity for carbon monoxide (DLCO; measuring gas exchange across the lung); maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) maneuvers (evaluating respiratory muscle strength); and impulse oscillometry (IOS; measuring lung mechanics). Each test will be performed at least 2-3 times to ensure the results are consistent. For all tests, the participant will breathe through a rubber mouthpiece with nose clips on to occlude the nasal passage.

Cardiopulmonary Exercise Tests: The participants will perform exercise on a stationary bicycle at each visit. While exercising, they will breathe through a mouthpiece with nose clips on, which allows for the breath-by-breath recording of physiologic variables throughout exercise. For each test, the participant will begin by sitting on the bike at rest (no pedaling) for approximately 6 minutes to establish a consistent measure of their baseline breathing. They will then begin pedaling for 1 minute against no resistance to warm-up. The load will then increase either by 10 Watts every minute (Visit 1) or to a constant work rate that will be maintained for 4 minutes (Visits 2-5). Every 2 minutes, the participant will be asked to take a full breath all the way in (an inspiratory capacity (IC) maneuver). The participant will also be asked to rate their breathing discomfort, their leg discomfort, how unpleasant their breathing feels, and how difficult it is to breathe in and out, using a 10-point Borg Scale.

Diaphragm EMG and Respiratory Pressure Measurements: Before exercise, a topical anaesthetic spray will be applied to the nasal passages and throat and a thin catheter (diameter 2 mm) will be inserted by experienced personnel through the nose down the throat and into the esophagus ("food tube") and top part of stomach. This catheter measures the electric activity (EMG) of the diaphragm, which provides useful information about the inspiratory drive to breathe. It also measures pressures in the esophagus within the chest as well as in the stomach, which gives useful information about the work of breathing and breathing mechanics.

Blood Sampling: Small samples of blood will be taken from the earlobe before exercise, at 2-minute intervals during exercise, and after exercise. The participant's earlobe will be warmed using a warm, damp cloth (ensuring adequate blood flow to the skin surface) throughout the baseline rest period and exercise. A very small puncture will be made using a lancet (similar to a very fine needle-tip), and blood will be collected in small glass tubes < 1mm in size. These samples will be analysed for their blood gas content (oxygen and carbon dioxide), variables needed to calculate dead space (the proportion of the lung unable to adequately participate in gas exchange).

Study design: This will be a single-centre, randomized, double-blind, placebo-controlled crossover study evaluating the effects of inhaled nitric oxide on the intensity of breathlessness and the physiological responses to a standardized exercise task. After giving written informed consent, participants will complete 5 visits, each conducted in the morning 2-7 days apart.

Visit 1 (Screening): The participants will have a detailed medical history taken and physical examination conducted by a study physician. The participants will also have their symptoms of COPD evaluated by standard written questionnaires [modified Medical Research Council (mMRC) dyspnea scale, Baseline Dyspnea Index (BDI), and COPD Assessment Test (CAT)]. These questionnaires will be explained to the participant by the study personnel and will be used to determine if the participants meet the criteria of having moderate-to-severe activity-related breathlessness. The participants will then undergo a series of pulmonary (lung) function tests at rest to determine lung function. Participants will complete a symptom-limited, incremental workload, cardiopulmonary exercise test on a stationary bicycle to determine their maximal work rate (Wmax). The participant will exercise on the bike for as long as they can, with the resistance increasing by 10 Watts every 1 min (see description above). Cardiac status will be monitored by 12-lead ECG. Heart rate, oxygen saturation (SpO2), and blood pressure will be monitored throughout exercise.

Visits 2 & 3 (Run-In): The participants will be familiarized with the 4-min standardized cycle exercise test and breathing apparatus that will be completed for the remaining visits. This cycle exercise test will be performed at a constant load. The initial resistance selected will be 75% of their maximum workload (Wmax; determined from exercise test in Visit 1) with adjustments to the load made as needed. The goal of the resulting 4-min exercise test is to have a standardized protocol that allows the participants to become sufficiently breathless to assess the potential therapeutic effect of nitric oxide while not being so intense as to prevent them from completing the test.

Visits 4 and 5 (Treatment): The participants will complete the 4-min cycle exercise test at the work rate established in Visits 2 and 3 while breathing from a gas mixture consisting of either 1) inhaled nitric oxide (800 ppm) or 2) placebo (room air), each on a background of room air (21% oxygen; remainder nitrogen). Tests at Visits 4 and 5 will include detailed measurements of diaphragm electric activity (EMG) and respiratory mechanical measurements. Blood samples will be collected as described above: before exercise, at 2-minute intervals throughout exercise, and at the end of exercise.

ELIGIBILITY:
Inclusion Criteria:

1. clinically stable as defined by stable hemodynamic status, optimized medical treatment, no changes in medication dosage or frequency of administration with no hospital admission in the preceeding 6 weeks
2. current or ex-smokers (>=20 pack-years)
3. male or female >45 years of age
4. mild COPD as defined by Medical Research Council dyspnea scale >=3 and post-bronchodilator FEV1 >=80% predicted and FEV1/FVC <0.7 and <LLN
5. ability to perform all study procedures and provide/sign informed consent

Exclusion Criteria:

1. women of childbearing age who are pregnant or trying to become pregnant
2. active cardiopulmonary disease or other comorbidities that could contribute to dyspnea and exercise limitation
3. important contraindications to clinical exercise testing, including inability to exercise because of neuromuscular or musculoskeletal disease(s)
4. use of daytime oxygen, or exercise-induced O2 desaturation to <80% on room air
5. body mass index (BMI) <18.5 or =>35.0 kg/m2
6. echocardiographic evidence of pulmonary hypertension
7. prior history of pulmonary thromboembolism or systemic vasculopathy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Dyspnea Intensity | At 4 minutes from start of exercise
  Primary objective is to measure perceptual (e.g. intensity of dyspnea and leg discomfort) responses at isotime (maximum exercise time achieved by all participants) during a standardized cardiopulmonary exercise testing (cycle ergometer).
Inspiratory neural drive | At 4 minutes from start of exercise
  Primary objective is to measure inspiratory neural drive (IND) by diaphragm activation (EMGdi/EMGdi max) at isotime (maximum exercise time achieved by all participants) during cardiopulmonary exercise testing (cycle ergometer).

SECONDARY OUTCOMES:
Lung volumes | At 4 minutes from start of exercise
  Secondary objective is to measure lung volumes at isotime (maximum exercise time achieved by all participants) during cardiopulmonary exercise testing (cycle ergometer).
Trans-diaphragmatic Pressure (Pdi) | At 4 minutes from start of exercise
  Secondary objective is to measure trans-diaphragmatic pressure (Pdi) at isotime (maximum exercise time achieved by all participants) during cardiopulmonary exercise testing (cycle ergometer).
Gastric Pressure (Pga) | At 4 minutes from start of exercise
  Secondary objective is to measure gastric pressure (Pga) at isotime (maximum exercise time achieved by all participants) during cardiopulmonary exercise testing (cycle ergometer).
Esophageal Pressure (Pes) | At 4 minutes from start of exercise
  Secondary objective is to measure esophageal pressure (Pes) at isotime (maximum exercise time achieved by all participants) during cardiopulmonary exercise testing (cycle ergometer).
Metabolic and gas exchange | At 4 minutes from start of exercise
  Secondary objective is to measure metabolic and gas exchage (earlobe blood samples analyzed for blood gas content) at isotime (maximum exercise time achieved by all participants) during cardiopulmonary exercise testing (cycle ergometer).

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, Principal Investigator — Queen's University, Respiratory Investigation Unit
Locations (1):
- Respiratory Investigation Unit, Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No